CLINICAL TRIAL: NCT02772341
Title: Evaluation of Halotherapy as Asthma Treatment in Children: a Randomized, Controlled, Double-blind Prospective Pilot Study
Brief Title: Evaluation of Halotherapy as Asthma Treatment in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 0059-12- RMB-CTIL
Record Dates: First submitted 2016-04-10; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Asthma
Keywords: Asthma; Halotherapy; Airway hyper-reactivity; Metacholine
MeSH Terms: conditions — Asthma | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Salt room with halogenerator (Active Comparator): Asthmatic patients sitting in a salt room with salt aerosol produced by a halogenerator.
  Interventions: Device: Salt room with halogenerator
- Salt room without halogenerator (Placebo Comparator): Asthmatic patients sitting in a salt room without salt aerosol
  Interventions: Other: Salt room without halogenerator

INTERVENTIONS:
Device: Salt room with halogenerator — Patients were assigned to 14 sessions (7 weeks, twice weekly, 45 minutes each treatment) sitting in a salt room with salt aerosol produced by a halogenerator (study group) or halotherapy without salt aerosol (placebo). Both the walls and the ceiling of the salt room are completely covered with ESCO-(European Salt Company) type certified-origin rock salt. The temperature (20-24°C) and humidity (44-60%) are at constant values. The halogenerator is located outside the salt room.
  Other Names: Treatment
  Arms: Salt room with halogenerator
Other: Salt room without halogenerator — Patients were assigned to 14 sessions (7 weeks, twice weekly, 45 minutes each treatment) sitting in a salt room without salt aerosol (placebo). Both the walls and the ceiling of the salt room are completely covered with ESCO-(European Salt Company) type certified-origin rock salt. The temperature (20-24°C) and humidity (44-60%) are at constant values.
  Other Names: Placebo
  Arms: Salt room without halogenerator

SUMMARY:
Background: Asthma is a chronic inflammatory disorder requiring intermittent or continuous anti-inflammatory therapy. Patients often turn to alternative treatments as complements or replacements to conventional treatments.

Aim: To evaluate the effect of salt room chambers (halotherapy) on bronchial hyper- responsiveness (BHR), fractional exhaled nitric oxide (FeNO), and quality of life in children with asthma.

Patients: Children aged 5-13 years with a clinical diagnosis of mild asthma not receiving anti-inflammatory therapy.

Methods: Randomized, double-blind, placebo-controlled study assessing the effect of salt room therapy on BHR, FeNO, spirometry and pediatric asthma quality of life questionnaire (PAQLQ). The treatment period lasted 7 weeks, 14 sessions with (treatment group) or without salt halogenerator.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disorder requiring intermittent or continuous anti-inflammatory therapy. Patients often turn to alternative treatments as complements or replacements to conventional treatments.

Our aim: To evaluate the effect of salt room chambers (halotherapy) on bronchial hyper - responsiveness (BHR), fractional exhaled nitric oxide (FeNO), and quality of life in children with asthma.

Patients: Children aged 5-13 years with a clinical diagnosis of mild asthma not receiving anti-inflammatory therapy.

Methods: Randomized, double-blind, placebo-controlled study assessing the effect of salt room therapy on BHR, FeNO, spirometry and pediatric asthma quality of life questionnaire (PAQLQ). The treatment period lasted 7 weeks, 14 sessions with (treatment group) or without salt halogenerator.

Visit 1: Written parental consent. Demographics, child's asthma/atopy history, and family history of asthma/atopy/smoking. The Pediatric asthma quality of life questionnaire (PAQLQ) by the patient/caregiver and the interviewer. Each patient performed spirometry, methacholine challenge test (MCT) and FeNO measurements. Following a positive MCT, patients were randomized to 14 sessions (7 weeks, twice weekly, 45 minutes each treatment) sitting in a salt room with salt aerosol produced by a halogenerator (study group) or halotherapy without salt aerosol (placebo). Both the walls and the ceiling of the salt room are completely covered with European Salt Company (ESCO) type certified-origin rock salt. The temperature (20-24°C) and humidity (44-60%) are at constant values. The halogenerator is located outside the salt room.

In the study group, dry sodium chloride (NaCl) particles (~20μm) were blown into the salt room while the blower was working without NaCl in the placebo group. The patients could not tell if dry salt aerosol was generated by halogenerator or not. The patients were instructed to use inhaled β2beta agonists as needed and to report any asthma exacerbation, use of medication or health care visit.

Visit 2: After seven weeks, each patient was re-evaluated by spirometry, MCT, FeNO, and PAQLQ.

ELIGIBILITY:
Inclusion Criteria:

* 5-13 years
* Mild asthma
* Positive methacholine challenge test (MCV, PC20-FEV1 <16mg/ml)

Exclusion Criteria:

* Any Chronic Lung Disease
* Febrile Illness in last 2 weeks
* FEV1 < 65% in study day
* Bronchodilators over the past 24 hours prior to each study
* Participation in any other clinical studies over the past 4 weeks
* Any acute illness on the day of the MCT,
* Anti-inflammatory treatment (inhaled corticosteroids or montelukast) over the previous two weeks before the MCT).
* Systemic corticosteroids in the two months prior to enrollment
* Emergency room (ER) visit or hospital admission following a respiratory illness during the 2-month period prior to enrollment.
* Previous halotherapy treatment.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Provocative concentration causing a 20% fall in the forced expiratory volume at one second (PC20-FEV1) as assessed by Methacholine Challenge Test | Study visit 1,2 (7 wks)

SECONDARY OUTCOMES:
Determination of exhaled Nitric Oxide in exhaled breath | Study visit study 1,2 (7 wks)
  Fractional Exhaled NO
Pulmonary function as assessed by spirometry | Study visit study 1,2 (7 wks)
  Spirometry
Quality of life of childhood asthma as assessed by the Standardized Pediatric Asthma Quality of Life Questionnaire (PAQLQ) | Study visit study 1,2 (7 wks)

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, Prof., Principal Investigator — Rambam Health Care Campus